CLINICAL TRIAL: NCT03953911
Title: Increasing HPV Vaccination Rates Via Educational Interventions in Schools Located Within Cedars-Sinai Catchment Areas
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adriana Vidal, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro54249
Record Dates: First submitted 2019-04-03; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Human Papilloma Virus; HPV Vaccination; Health Education
MeSH Terms: conditions — Health Education | interventions — Mobile Health Units

STUDY DESIGN:
Intervention Model Description: In this parallel study, three middle schools located in Los Angeles County will be assigned to 2 intervention arms: control (mobile clinic-only every 6-months); intervention (mobile clinic every 6-months or every month PLUS weekly educational sessions for parents).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants at the Schools, providers of the mobile clinic and the outcomes assessor will be masked from the allocation of participants to the arms to ensure reduction in bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Mobile Clinic Only (Active Comparator): The middle school assigned to the control arm will receive a visit by a mobile clinic every 6 months only. The school will follow normal protocol for HPV vaccination awareness. Parents will be made aware of the mobile clinic per normal school newsletters and mailers.
  Interventions: Biological: Mobile Clinic
- Mobile Clinic plus Educational Sessions (Experimental): The middle school assigned to the Mobile Clinic every 6-mos or month plus Educational Sessions arm will receive visitation of a mobile clinic providing free HPV vaccination among other school-related vaccines once every 6-months or once a month. Parents will be made aware of the mobile clinic per normal school newsletters and mailers. In addition, parents will be provided with free weekly educational sessions about the HPV Vaccine as a cancer-prevention effort.
  Interventions: Biological: Mobile Clinic; Behavioral: Educational Sessions for Parents

INTERVENTIONS:
Biological: Mobile Clinic — This intervention involves the availability of a free mobile clinic operated by Cedar-Sinai Medical Center providing free HPV vaccinations at school campuses.
Behavioral: Educational Sessions for Parents — This intervention involves providing free weekly educational sessions for parents of students at the participant schools pertaining to the HPV Vaccination.
  Arms: Mobile Clinic plus Educational Sessions

SUMMARY:
Infections with human papillomavirus (HPV) can cause cancer of the cervix, vagina, anus, throat, mouth, and penis. Prevention of these HPV-related cancers could be achieved by immunization with the nonavalent (HPV6,11,16,18,31,33,45,52,58) vaccine currently commercially available. However, in the U.S. approximately only 30% of females and 20% of males in the recommended age group receive the complete, three-dose HPV vaccine. Furthermore, data from the Los Angeles county suggest that HPV vaccination rates among these groups are lower than the national average. Significant barriers clearly remain including knowledge of the vaccine, transportation, number of doses and concern of side effects. Several programs worldwide have shown that schools remain an important venue for education as well as vaccination. In the US, vaccination within schools remains difficult because of many barriers including lack of nursing, insurance reimbursement, and liability. However, the school remains an important access to educational formats. The objective of this study is to evaluate the effectiveness of educational sessions on the HPV vaccine among parents with children of vaccination age as a strategy to increase HPV vaccine uptake, by comparing HPV vaccination rates before and after the intervention. It is hypothesized HPV vaccine uptake will improve through the receipt of educational sessions to the parents of middle school children about the importance of the anti-cancer vaccine, the HPV vaccine. Three schools within Cedars-Sinai catchment area with whom Cedars-Sinai already has a Memorandum of Understanding in place: Berendo, Drew, and Carver Middle Schools in Los Angeles (SPA 4, SPA 6) will be recruited to the study. HPV vaccination rates will be compared before and after the intervention at the end of the observation period (12 months).

DETAILED DESCRIPTION:
Rationale and Significance

Infections with human papillomavirus (HPV) can cause cancer of the cervix, vagina, anus, throat, mouth, and penis. Prevention of these HPV-related cancers could be achieved by immunization with the nonavalent (HPV6,11,16,18,31,33,45,52,58) vaccine currently commercially available. However, in the U.S. approximately only 30% of females and 20% of males in the recommended age group receive the complete, three-dose HPV vaccine. The vaccine is covered under Vaccine for Children Program so the underinsured and uninsured have access. Furthermore, data from the Los Angeles county suggest that HPV vaccination rates among these groups are lower than the national average. Significant barriers clearly remain including knowledge of the vaccine, transportation, number of doses and concern of side effects. Several programs worldwide have shown that schools remain an important venue for education as well as vaccination. In the US, vaccination within schools remains difficult because of many barriers including lack of nursing, insurance reimbursement, and liability. However, the school remain an important access to educational formats. Barriers associated with the HPV vaccine uptake is the initial stigmatizing information created by anti-vaccine groups, providers not recommending the vaccine and not understanding the cancer prevention strategies (i.e. getting vaccination prior to exposure).

Barriers to HPV vaccination

Although the US has invested in a large national effort toward improvement of HPV vaccination rates, little progress has been achieved since 2006. While financial access should not be a barrier to vaccination for most children, some insurance plans do not cover vaccines. Several factors appear to influence vaccination rates: a) limited understanding of HPV and HPV-related diseases by parents and patients; b) parental safety concerns about the vaccine; c) provider discomfort talking about sexual behavior; d) providers lack of time for discussions about the vaccine; e) parental perception that there is no clear recommendation from a health care provider; f) parental belief that son or daughter is too young for the vaccine because they are not sexually active; and g) provider concern that there is lack of adequate reimbursement. In LA County, lack of knowledge that a cancer vaccine exists, lack of transportation, and fear of immigration status disclosure are further barriers to vaccination.

We hypothesize HPV vaccine uptake will be improved through the receipt of educational sessions to the parents of middle school children about the importance of the anti-cancer vaccine, the HPV vaccine.

Such sessions will increase knowledge about HPV vaccine availability, as well as improve the perceptions around HPV vaccination. Vaccination rates are lower in the Service Planning areas (SPA) 4 and 6 compared to SAP 5 (West LA).

Primary Objectives

To evaluate the ability of educational sessions about the HPV vaccine to increase HPV vaccine uptake, by comparing HPV vaccination rates before and after the intervention.

Endpoints

The primary outcome will be HPV vaccination rates. Vaccination rates will be compared between before (baseline) and after the intervention at the end of the observation period (12 months). We expect to find higher HPV vaccine rates after the intervention.

Study Design

We will recruit 3 schools within Cedars-Sinai catchment area with whom Cedars-Sinai already has a Memorandum of Understanding in place: Berendo, Drew, and Carver Middle Schools in Los Angeles (SPA 4, SPA 6). These MOUs were obtained through the Cedars-Sinai Coach-for Kids Program Director, Michele Rigsby-Pauley, a co-investigator in this study. We will first conduct focus group interviews with parents to learn about parents' concerns about the HPV vaccine and to identify important messages for parents. These would also include strategies for dissemination of information (PTA meetings, text messages to parents, online education). HPV vaccination rates will be compared before and after the intervention at the end of the observation period (12 months).

ELIGIBILITY:
Inclusion Criteria:

* age 11-13
* student of a participating middle school assigned to Arm 2 or Arm 3

Exclusion Criteria:

* already received the HPV vaccine

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2019-05-28 (Estimated); Primary Completion 2020-05-27 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination rates | 12 months
  The primary outcome will be HPV-vaccination rates. Vaccination rates will be compared between baseline and intervention (12 months) between the intervention and control arms. We will conduct at least 50 educational sessions. Briefly, using a two-sided Z-test with unpooled variances with 5% significance.

IPD SHARING:
Plan to Share IPD: No